CLINICAL TRIAL: NCT02078999
Title: Observational Study in Patients Admitted in the Intensive Care Unit.Tracheal Bacterial Load Surveillance in Patients Undergoing Mechanical Ventilation - Assessment of Biomarkers in the Distinction Between Colonization and Infection
Brief Title: Biomarkers in Patients Undergoing Mechanical Ventilation
Acronym: VAP
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Hospital Universitari Vall d'Hebron Research Institute (Other); Hospital Clinic of Barcelona (Other); Centro Hospitalar Lisboa Ocidental (Other Government); Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Antonio Artigas Raventós, PhD, Corporacion Parc Tauli
Other Study IDs: Ventilator-adquired Pneumonia; VAP2008 (Other: Parc Tauli IRB)
Record Dates: First submitted 2012-08-03; First posted 2014-03-05 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Ventilator Associated Pneumonia
Keywords: Mechanical ventilation, procalcitonin, c-reactive protein
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bronchoalveolar lavage,biochemical lab,exhaled air.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Control Grup: * Daily clinical data collection
  * Quantitative tracheal aspirates (QTA) every 3 days
  * Deep freeze serum samples for posterior analysis every day (two aliquots).
  * In patients with documented pneumonia daily collection of the following variables will continue: CRP, PCT, ABG, mechanical ventilation parameters, ACCP/SCCM consensus conference criteria, simplified CPIS, SOFA.
- Patients with pulmonary infection: * Daily clinical data collection
  * Quantitative tracheal aspirates (QTA) every 3 days
  * Deep freeze serum samples for posterior analysis every day (two aliquots).
  * In patients with documented pneumonia daily collection of the following variables will continue: CRP, PCT, ABG, mechanical ventilation parameters, ACCP/SCCM consensus conference criteria, simplified CPIS, SOFA.
- Patients with extrapulmonary infection: * Daily clinical data collection
  * Quantitative tracheal aspirates (QTA) every 3 days
  * Deep freeze serum samples for posterior analysis every day (two aliquots).
  * In patients with documented pneumonia daily collection of the following variables will continue: CRP, PCT, ABG, mechanical ventilation parameters, ACCP/SCCM consensus conference criteria, simplified CPIS, SOFA.

SUMMARY:
To evaluate in a cohort of patients on mechanical ventilation, for non-infectious reasons and for documented sepsis of pulmonary as well as non-pulmonary origin, the bacterial load, procalcitonine (PCT), C-Reactive Protein (CRP), temperature, White cell count (WCC), American College of Chest Physicians/Society of Critical Care Medicine (ACCP/SCCM) consensus conference criteria, Sequential Organ Failure Assessment score (SOFA) and simplified Clinical Pulmonary Infection Score (CPIS) through the mechanical ventilation period

DETAILED DESCRIPTION:
The investigators hypotized that:

1. In patients on mechanical ventilation for a non-infectious cause of respiratory failure, the tracheal bacterial load should be absent or below the cut-off values defined for infection, that is to say tracheal colonization.
2. In patients without the diagnosis of Ventilator-Adquired Pneumonia (VAP) and not taking antibiotics till the weaning process, tracheal bacterial load should remain below the predefined cut-off values and the biomarkers (PCT and CRP) should be surrogate markers of this clinical course.
3. In patients developing VAP, an increase in tracheal bacterial load should precede diagnosis with an associated rise in the biomarkers levels (PCT and CRP). Finally, after institution of antibiotic therapy, adequate therapy should be associated with a decrease tracheal bacterial load as well as of the biomarkers (PCT and CRP).
4. In patients admitted with clinical suspicion of pneumonia, either community-acquired (CAP) or hospital-acquired (HAP), with microbiological documentation, after institution of antibiotic therapy, adequate therapy should be associated with a decrease tracheal bacterial load as well as the biomarkers (PCT and CRP).
5. In patients admitted with clinical suspicion of a non-pulmonary infection (e.g. peritonitis and urosepsis) and on mechanical ventilation for an expected length longer than 3 days, either community or hospital-acquired, preferentially with microbiological documentation, after institution of antibiotic therapy, adequate therapy should be associated with a decrease of biomarkers (PCT and CRP).

ELIGIBILITY:
Inclusion criteria:

* Patients admitted in the ICU, with an expected length of mechanical ventilation > 3 days.
* Not receiving antibiotics for >24 hrs before ICU admission- An expected length of mechanical ventilation > 3 days

Exclusion Criteria:

* Patients <18 yrs old
* Pregnancy and lactation
* Fulminant hepatic failure
* Pancreatitis
* Patients with the diagnosis of disseminated cancer, expected to die or undergo withdrawal of treatment within 72 hours after enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in the ICU
Sampling Method: Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Procalcitonine (PCT) levels evolution | Up to 21 days
  Procalcitonin (PCT) levels assessed daily up to 21 days

SECONDARY OUTCOMES:
C-Reactive Protein (CRP) | Up to 21 days
  To evaluate the value of serum C-Reactive Protein (CRP) concentrations in the distinction between colonization and pulmonary infection
Biomarkers at day of Ventilator-Adquired Pneumonia (VAP) | Up to 21 days
  Measurement of biomarkers namely, copeptin, adrenomedulin, atrial natriuretic peptide, Interleukine 6, Interleukine 1 and hydrogen peroxide

CONTACTS AND LOCATIONS:
Overall Officials: torres antonio, doctor, Principal Investigator — hospital vall hebron barcelona; palomar mercedes, doctor, Principal Investigator — Hospital Clinic i provincial de Barcelona; povoa pedro, doctor, Principal Investigator — Centro hospitalario de lisboa occidental
Locations (1):
- Hospital Parc Taulí, Sabadell, Barcelona, Spain

REFERENCES:
- [Result] Povoa P, Martin-Loeches I, Ramirez P, Bos LD, Esperatti M, Silvestre J, Gili G, Goma G, Berlanga E, Espasa M, Goncalves E, Torres A, Artigas A. Biomarker kinetics in the prediction of VAP diagnosis: results from the BioVAP study. Ann Intensive Care. 2016 Dec;6(1):32. doi: 10.1186/s13613-016-0134-8. Epub 2016 Apr 14. PMID 27076187
- [Result] Martin-Loeches I, Bos LD, Povoa P, Ramirez P, Schultz MJ, Torres A, Artigas A. Tumor necrosis factor receptor 1 (TNFRI) for ventilator-associated pneumonia diagnosis by cytokine multiplex analysis. Intensive Care Med Exp. 2015 Dec;3(1):26. doi: 10.1186/s40635-015-0062-1. Epub 2015 Sep 16. PMID 26377207
- [Derived] Ceccato A, Camprubi-Rimblas M, Bos LDJ, Povoa P, Martin-Loeches I, Forne C, Areny-Balaguero A, Campana-Duel E, Morales-Quinteros L, Quero S, Ramirez P, Esperatti M, Torres A, Blanch L, Artigas A. Evaluation of the Kinetics of Pancreatic Stone Protein as a Predictor of Ventilator-Associated Pneumonia. Biomedicines. 2023 Sep 29;11(10):2676. doi: 10.3390/biomedicines11102676. PMID 37893050
- [Derived] Povoa P, Martin-Loeches I, Ramirez P, Bos LD, Esperatti M, Silvestre J, Gili G, Goma G, Berlanga E, Espasa M, Goncalves E, Torres A, Artigas A. Biomarkers kinetics in the assessment of ventilator-associated pneumonia response to antibiotics - results from the BioVAP study. J Crit Care. 2017 Oct;41:91-97. doi: 10.1016/j.jcrc.2017.05.007. Epub 2017 May 8. PMID 28502892